CLINICAL TRIAL: NCT03599115
Title: The Effects of Food-Specific Inhibitory Control Training on Weight, Diet, and Neural Indices in Overweight and Obese Adults
Brief Title: Effects of Inhibitory Control Training in Eating Behaviors
Acronym: N2ICT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham Young University (Other)
Responsible Party: Principal Investigator, Kaylie Carbine, Principal Investigator, Brigham Young University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: X17021
Record Dates: First submitted 2018-06-25; First posted 2018-07-26 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Overweight and Obesity
Keywords: inhibitory control training; food; event-related potentials; weight reduction
MeSH Terms: conditions — Overweight; Obesity; Weight Loss

STUDY DESIGN:
Intervention Model Description: There are two arms of this study: food-specific inhibitory control training (condition of interest) and a generic inhibitory control training (active control). Given baseline levels of inhibitory control (assessed at baseline visit), participants are randomly assigned to the generic or food-specific month long inhibitory control training. All other protocols, including baseline and follow-up visits and assessment of food intake and weight, are identical and follow the same time line across the two arms.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants are told there is only one intervention for the study and are not aware if they have been assigned to the intervention group or the active control. Research assistants collecting data are blind to what arm the participant was assigned to. During data preprocessing steps, individuals will be blind to what group a participant belongs too (and all data will be preprocessed together). Only when conducting statistical analyses will the principle investigator be aware of what participant belongs to what group, in order to conduct group analyses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inhibitory Control Training to Food Items (Experimental): Participants complete a 10 minute training task once a day, 4 days a week, for 4 weeks. Task is administered using a mobile app (Paradigm mobile) that is installed on an iPhone or iPad. Participants receive an instruction text/email at 9am on their chosen weekdays with instructions on what task to complete and a reminder text/email at 5pm if the task has not yet been completed. Research team receives an email when the task has been completed. When the task is administered, participants see a picture for 1250ms with an inter-stimulus interval of 1250ms and have to indicate which side of the screen the picture appears (go trials). Participants are instructed to not make a response when the picture is surrounded by a black box (no-go trials). There are 6 blocks with 36 trials each, half being go and half being no-go trials. High-calorie foods are always no-go trials and low-calorie foods are always go trials.
  Interventions: Behavioral: Inhibitory Control Training
- Inhibitory Control Training to Neutral Items (Active Comparator): Participants complete a 10 minute training task once a day, 4 days a week, for 4 weeks. Task is administered using a mobile app (Paradigm mobile) that is installed on an iPhone or iPad. Participants receive an instruction text/email at 9am on their chosen weekdays with instructions on what task to complete and a reminder text/email at 5pm if the task has not yet been completed. Research team receives an email when the task has been completed. When the task is administered, participants see a picture for 1250ms with an inter-stimulus interval of 1250ms and have to indicate which side of the screen the picture appears (go trials). Participants are instructed to not make a response when the picture is surrounded by a black box (no-go trials). There are 6 blocks with 36 trials each, half being go and half being no-go trials. All pictures are of household items.
  Interventions: Behavioral: Inhibitory Control Training

INTERVENTIONS:
Behavioral: Inhibitory Control Training — Computerized go/no-go task where individuals make responses to certain items (go trials) and withhold responses from certain items (no-go trials, in this case, trials surrounded by a black box). Intervention is designed to target and improve inhibitory control cognitive mechanisms in general (generic arm) or towards high-calorie foods specifically (food arm).

SUMMARY:
Overweight and obese individuals will be randomly assigned to a food-specific or generic inhibitory control training. Food intake, weight, and neural indices of inhibitory control will be assessed prior, immediately after the 4-week intervention, and 12-weeks after intervention completion to assess the effectiveness of a mobile inhibitory control training intervention over time for health outcomes.

DETAILED DESCRIPTION:
All participants will report to the lab for a baseline session, where their weight, average food intake for three days (using the Automated Self-Administer 24-hour Dietary Recall [ASA24] system), neural indices of inhibitory control (as assessed by the N2 event-related potential component during a food and genetic go/no-go task), appetitive drive toward food (as measured by the Power of Food Scale) and basic demographic information will be assessed. Based off their gender and baseline levels of inhibitory control (indicated by the N2), participants will be assigned to a four week food-specific inhibitory control training or a generic inhibitory control training. Trainings are administered on a mobile device via an app and participants select four our of five business days to complete the trainings on. Immediately after the four weeks, participants will come in for a follow-up session where their weight, food intake, N2, and appetitive drive to food will be assessed again. Finally, participants will have a 12-week waiting period where they do not complete the trainings. After the 12 weeks, they will come in for a final lab visit where their weight, food intake, N2, and appetitive drive to food will be assessed one last time.

ELIGIBILITY:
Inclusion Criteria:

* Overweight or Obese (BMI > 25 kg/m2)

Exclusion Criteria:

* Diagnosis of a psychological disorder (e.g., major depressive disorder, general anxiety disorder), neurological disorder (e.g., epilepsy, stroke), learning disability, or eating disorder (e.g., anorexia nervosa, bulimia nervosa, binge eating disorder)
* Metabolic/chronic disease (e.g., cardiovascular disease, Type II diabetes)
* Pregnant or lactating
* Current participation in a weight loss diet
* Food allergies
* Head injury that resulted in a loss of consciousness
* Avid exercisers (i.e., participate in at least 20 minutes of vigorous physical activity more than three times a week)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 2017-09-26 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Caloric Intake | Three days will be completed at baseline, immediately after the intervention, and at the 12 week follow-up visit (total of 9 recalls)
  Using the Automated Self-Administered 24-hour Dietary Recall (ASA24), participants will record their food intake for two weekdays and one weekend, two of which will be randomly assigned and one which will be the day they report to their lab visit. Caloric intake, as quantified by ASA24, will be averaged for the three days and statistically analyzed to see if average caloric intake changes over time due to the inhibitory control training arm.
Weight | Assessed at baseline, immediately after the intervention, and at the 12-week follow-up visit.
  Weight will be measured in kilograms using a stadiometer to see if weight changes over the course of the study.
N2 Event-Related Potential Component | Assessed at baseline, immediately after the intervention, and at the 12-week follow-up visit.
  The N2 is a negative deflection in the event-related potential waveform occurring 200 to 300 ms after the onset of a stimulus and is larger (i.e., more negative) when an individual has to withhold a dominant response. It is a neural reflection of inhibitory control. The investigators will assess if the N2 amplitude gets larger as a result of inhibitory control training (as individuals will be better at recruiting inhibitory control resources). The investigators will also see if the N2 predicts who is successful at losing weight and reducing caloric intake after the intervention, to better understand the mechanism of action for inhibitory control training.

SECONDARY OUTCOMES:
No-Go Accuracy | Assessed at baseline, immediately after the intervention, and at the 12-week follow-up visit.
  Percent of correct no-go trials during the laboratory go/no-go tasks. The investigators are interested if this improves due to the intervention.
Correct Go Reaction Times | Assessed at baseline, immediately after the intervention, and at the 12-week follow-up visit.
  Time in ms to correctly respond to a go trial during the laboratory tasks. The investigators are interested if reaction times get faster due to the intervention.

OTHER OUTCOMES:
Power of Food Scale (PFS) | Assessed at baseline, immediately after the intervention, and at the 12-week follow-up visit.
  The PFS assesses thoughts, feelings, and motivations to consume palatable food. It provides a measure of the appetitive drive individuals have to consume food. There are 15 items on the PFS, each ranging from 1 (don't agree at all) to 5 (strongly agree). The PFS is divided into 3 subscales that assess appetitive drive in 3 different environmental situations: when food is available (6 items), when food is physically present (4 items), and when food has been tasted (5 items). Subtotal scores are calculated by taking the mean of all the individual items in each subscale (subscale scores ranging from 1 to 5). An overall score, which is calculated by averaging the three subscale scores, will be used as the outcome of interest (overall score ranging from 1 to 5). A higher overall score on the PFS indicates there is a higher appetitive drive to consume food. The investigators will test if the appetitive drive to consume food changes over time due to the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham Young University, Provo, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
Study protocol, materials, and analysis plans are already posted on the Open Science Framework (https://osf.io/szxua/). Actual study data (de-identified) will be made available, along with analysis codes, once the study has been complete and published.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Once data collection and data analysis has been completed and published in a scientific journal, the study data (de-identified) will either be posted on an open science website, such as the Open Science Framework, or will be given to other researchers upon request.
URL: https://osf.io/szxua/

REFERENCES:
- See also: Open Science Framework study specific page — https://osf.io/szxua/